CLINICAL TRIAL: NCT06076668
Title: Dexmedetomidine Infusion Versus Oral Melatonin for Prevention of Intensive Care Unit (ICU) Delirium; A Prospective Randomized Controlled Study
Brief Title: Dexmedetomidine Infusion Versus Oral Melatonin for Prevention of Intensive Care Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, eslam salem, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmedetomidine
Record Dates: First submitted 2023-09-16; First posted 2023-10-11 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Dexmedetomidine; Melatonin; Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Melatonin; Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D (n=30) (Experimental): patients will receive intravenous dexmedetomidine infusion of 0.2 mcg/kg/h starting at 9 p.m. The infusion will be halved at 6:00 A.M. and discontinued at 6:15 A.M.
  Interventions: Drug: Dexmedetomidine
- Group M (n=30) (Experimental): patients will receive oral melatonin tablet 3 mg at 9:00 p.m.
  Interventions: Drug: Melatonin 3 MG
- Control group (Placebo Comparator): patients will receive saline infusion at the same rate of dexmedetomidine infusion and placebo capsule similar to that of melatonin.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive an intravenous dexmedetomidine infusion of 0.2 mcg/kg/h starting at 9 p.m. The infusion will be halved at 6:00 A.M. and discontinued at 6:15 A.M.
  Other Names: DEX group
  Arms: Group D (n=30)
Drug: Melatonin 3 MG — Patients will receive oral melatonin tablet 3 mg 9:00 p.m.
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: Group M (n=30)
Drug: Saline — Patients will receive saline infusion at the same rate of dexmedetomidine infusion and placebo capsule similar to that of melatonin.
  Other Names: Control group
  Arms: Control group

SUMMARY:
This study aims to compare the effect of dexmedetomidine infusion and oral melatonin on preventing delirium in intensive care unit (ICU) patients.

DETAILED DESCRIPTION:
Delirium is experienced in 20% to 40% of the critically ill and up to 80% of mechanically ventilated (MV) medical or surgical patients . It is a confessional state that has been described as a transient global disorder of cognition, awareness, and attention and as such is not only challenging for the treating medical team, but also has a considerable impact on affected patients. It is associated with prolonged hospital length of stay and time on MV, deterioration in cognition, and increased morbidity and mortality causing additional health-care expenses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years or older.
* Either gender.
* Healthy gastrointestinal function (patients tolerated oral medications by gavage or mouth).
* Richmond Agitation Sedation Scale (RASS) >-1.
* No basic delirium or mood changes before admission to intensive care unit(ICU).

Exclusion Criteria:

* Patient refusal.
* History of irreversible brain disease consistent with severe dementia.
* Patient admitted with a primary neurologic condition or injury (e.g., intracranial hemorrhage).
* Heart rate (HR) less than 50 beats/ min or second- third degree heart block in the absence of a pacemaker.
* Acute alcohol withdrawal requiring benzodiazepine administration.
* History of hepatic encephalopathy or end-stage liver disease (Child-Pugh class B or C).
* The expected duration of intensive care unit (ICU) stay less than 5 days.
* Inability to obtain informed consent.
* Pregnancy.
* Allergy to dexmedetomidine or melatonin.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of delirium | 14 days from admission to intensive care unit
  The incidence of delirium within 14 days from admission to the intensive care unit (ICU) or until ICU discharge before this time. Every 12 hours throughout the study.

SECONDARY OUTCOMES:
The onset of delirium. • Duration of delirium. • Frequency of delirium. • Length of ICU stay. • Total dose of Haloperidol per day. | 14 days from admission to intensive care unit
  Delirium was assessed using Confusion Assessment Method for intensive care unit (CAM- ICU) score at admission to ICU and every 12hr throughout the study.
  The final CAM-ICU score ranges from 0-7 with 7 being most severe. CAM-ICU-7 scores were further categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Duration of delirium | 14 days from admission to intensive care unit
  Delirium was assessed using Confusion Assessment Method for intensive care unit(CAM- ICU) score at admission to ICU and every 12hr throughout the study.
  The final CAM-ICU score ranges from 0-7 with 7 being most severe. CAM-ICU-7 scores were further categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Frequency of delirium | 14 days from admission to intensive care unit
  Delirium was assessed using Confusion Assessment Method for intensive care unit(CAM- ICU)score at admission to ICU and every 12hr throughout the study.
  The final CAM-ICU score ranges from 0-7 with 7 being most severe. CAM-ICU-7 scores were further categorized as 0-2: no delirium, 3-5: mild to moderate delirium, and 6-7: severe delirium.
Total dose of Haloperidol per day | 14 days from admission to intensive care unit
  Total dose of Haloperidol per day 14 days from admission to intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.